CLINICAL TRIAL: NCT06017414
Title: Systemic Psychotherapy-informed Self-help and Paraprofessional Training in a Naturalistic Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gunther Meinlschmidt (Other)
Responsible Party: Sponsor-Investigator, Gunther Meinlschmidt, Prof. Dr., International Psychoanalytic University Berlin
Organization: International Psychoanalytic University Berlin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IPU_ST_2023_05
Record Dates: First submitted 2023-08-22; First posted 2023-08-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Psychological Distress
Keywords: Psychological Distress; Emotional Distress; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Intervention Model Description: Our study is comprised of two main components:
  An exploratory randomized, natural setting, pre-post-follow-up study design based on systemic principles and techniques assessing changes over time, and comparing:
  1. the OSI/growth path training condition with a waitlist comparator condition,
  2. paraprofessional provider/listener training condition with a waitlist comparator condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Growth Path Intervention (Experimental): Participants for this arm are members of the 7 Cups platform (signed up as 'members', but not signed up as 'listeners') who will receive the Systemic Psychotherapy-informed growth path intervention.
  Interventions: Behavioral: Systemic Psychotherapy-informed Growth Path
- Waitlist followed by Growth Path Intervention (No Intervention): Participants for this arm are members of the 7 Cups platform (signed up as 'members', but not signed up as 'listeners'). The waitlist comparator condition has 7 Cups access and use as usual during the waitlist period. Participants will receive access to the Systemic Psychotherapy-informed growth path intervention after the waitlist condition of 7 weeks is completed.
- Listener Training Intervention (Experimental): Participants for this arm are listeners on the 7 Cups platform (signed up as 'listeners', but not signed up as 'members') who will receive the Systemic Psychotherapy-informed listener training intervention.
  Interventions: Behavioral: Systemic Psychotherapy-informed Listener Training
- Waitlist followed by Listener Training Intervention (No Intervention): Participants for this arm are listeners on the 7 Cups platform (signed up as 'listeners', but not signed up as 'members'). The waitlist comparator condition has 7 Cups access and use as usual during the waitlist period. Participants will receive access to the Systemic Psychotherapy-informed listener training intervention after the waitlist condition of 7 weeks is completed.

INTERVENTIONS:
Behavioral: Systemic Psychotherapy-informed Growth Path — A self-guided program lasting 5 weeks on the 7 Cups platform. The self-help intervention aims to support members to explore their relationships, situations, and goals.
  Arms: Growth Path Intervention
Behavioral: Systemic Psychotherapy-informed Listener Training — A self-guided program lasting 5 weeks on the 7 Cups platform. The self-help intervention encourages listeners to explore their relationships, situations, and goals and think about how they would support members working through their own relationships, situations, and goals.
  Arms: Listener Training Intervention

SUMMARY:
The main goal of this project is to address several gaps in the current literature in an exploratory way, by generating data via a synthesized research design. There are three fields of research this project seeks to have a meaningful impact on: the digital implementation of systemic psychotherapy-informed principles and approaches into unguided self-help growth paths, the training of paraprofessional mental health service providers with systemic psychotherapy-informed listener training, and the utilization of paraprofessional mental health service providers in the delivery of online guided systemic psychotherapy-informed self-help interventions.

This impact will be derived from addressing the following research questions:

* Are online self-help interventions based on systemic psychotherapy approaches and principles feasible?
* Are online self-help interventions based on systemic psychotherapy approaches and principles efficacious (as compared to a waitlist), indicated by mental-health-related outcomes of participants?
* Is training of paraprofessionals in guiding the use of self-help interventions based on systemic psychotherapy approaches and principles feasible?
* Is this training of paraprofessionals based on systemic psychotherapy approaches and principles efficacious (as compared to a waitlist), indicated by mental-health-related outcomes of trainees?

DETAILED DESCRIPTION:
A comprehensive systematic review was published showing the efficacy and effectiveness of Systemic Psychotherapy in treating the most common psychological disorders. It is important to critically evaluate Systemic Psychotherapy to identify the most promising paths forward. One such promising path lies in online self-help interventions (OSIs). OSIs can be broadly divided into guided and unguided modes of self-help, with the former showing better efficacy than the latter. This distinction notwithstanding, unguided OSIs have been shown to be effective in the treatment of anxiety, depression, the prevention of suicides, and numerous other psychological disorders and conditions. From a public health perspective, OSIs are particularly interesting as they promise to address several obstacles to conventional mental health care provision and harness patients' capacities for self-help. Additionally, their scalability might facilitate the provision of services to target groups that could otherwise not be reached. Platforms such as "7 Cups" (https://www.7cups.com), which provides OSIs (called Growth Paths), text-based paraprofessional peer support, paraprofessional training (called Listener Training), and signposting to professional services, have been identified as particularly effective in incorporating this approach. Platforms such as 7 Cups, whose peer support programme has received some attention, warrant further scrutiny. While it is acknowledged as an important part of improving access to mental health care globally, there is only one published study on an OSI explicitly incorporating methods and techniques associated with Systemic Psychotherapy and no studies examining paraprofessional training in a widely accessible online platform such as 7 Cups. This exploratory study aims to make a timely and meaningful contribution towards the gaps in the current literature.

ELIGIBILITY:
Inclusion Criteria:

* Have been signed up on the 7Cups platform as a member or listener for a minimum of 3 months.
* The intended 7Cups member is "anyone who wants to talk about whatever is on their mind" and the intended 7Cups listener is anyone who does the basic training and "wants to listen to members" (https://www.7cups.com/about/), including given consent to data use.
* Have actively used the 7Cups platform as a member or listener by logging into the platform at least once in the last 2 weeks.
* Agree to participate in our study and provide consent to data usage.
* Aged 18 years or above.
* English language (sufficient capacity to interact with the 7Cups platform and participate in the assessments).

Exclusion Criteria:

* Refusal to consent with data use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale 6 (K6) (Short version of the K10) (Cornelius et al., 2013; Kessler et al., 2002). | Intervention condition is measured before, directly after, and 2 weeks after the 5 week intervention. Waitlist condition is measured at parallel timepoints, then receives the intervention and follows the intervention condition measurement time frame.
  The K6 is a standardized self-reported outcome assessment tool used to measure global non-specific psychological distress with questions relating to depressive and anxiety symptoms. The K6 consists of 6 items asking people to rate their emotional states on a 5-point Likert scale ranging from ''All the time'' to ''None of the time''. Scores are summed and yield a score of 0 to 24. Higher scores indicate increased non-specified psychological distress.

SECONDARY OUTCOMES:
Perceived Stress Scale 4 (PSS-4) (Short version of the PSS-10) (Warttig et al., 2013). | Intervention condition is measured before, directly after, and 2 weeks after the 5 week intervention. Waitlist condition is measured at parallel timepoints, then receives the intervention and follows the intervention condition measurement time frame.
  The PSS-4 is a standardized patient-reported outcome assessment tool used to measure global perceptions of stress from the individual's perspective. The PSS-4 consists of 4 items asking people to evaluate their experience of stressful situations on a 5-point Likert scale ranging from 'never' to 'very often'. Scores are summed and yield a score of 0 to 16. The higher the score on the PSS-4, the greater the person evaluates that the stressful situations are beyond their ability to deal with them.
Patient Health Questionnaire (PHQ-4) (Kroenke, Spitzer, & Williams, 2003). | Intervention condition is measured before, directly after, and 2 weeks after the 5 week intervention. Waitlist condition is measured at parallel timepoints, then receives the intervention and follows the intervention condition measurement time frame.
  The PHQ-4 consists of the first two items of the PHQ-9 and GAD-7, respectively. This comprises the two principal DSM items for major depressive disorder and generalized anxiety disorder, respectively. Each ranges from a score of 0 to 6. The PHQ-4 uses a on a 4-point Likert scale ranging from 'not at all' to 'nearly every day'. Higher scores indicate higher levels of depressive and anxiety symptoms.
Multidimensional Mood State Questionnaire (MDMQ, good-bad subscale) (English-language version of MDBF) (Steyer, Schwenkmezger, Notz, & Eid, 1997). | Intervention condition is measured before, directly after, and 2 weeks after the 5 week intervention. Waitlist condition is measured at parallel timepoints, then receives the intervention and follows the intervention condition measurement time frame.
  The MDBF measures participant current mood (good-bad). The MDBF uses a 6-point Likert scale ranging from 'definitely not' to 'extremely'. Scores are summed, yielding a total score of 4 to 24. Higher scores indicate higher good mood scores.

OTHER OUTCOMES:
Usability Metric for User Experience Questionnaire (UMUX-LITE) (Finstad, 2010) | Intervention condition is measured after the 5 week intervention (Intervention condition only).
  Assesses the Usability of the intervention delivery. The UMUX-LITE uses a 7-point Likert scale. Item responses are recoded to compute a score ranging from 0 to 100. Higher scores indicate increased ratings of the system's capabilities and ease of use.
Qualitative questionnaire. | Intervention condition is measured after the 5 week intervention (Intervention condition only).
  By using Revicki (2003), Ghani (2015) and Johnson et al. (2011) as guidance a set of questions were designed to get further information and details about the experience and quality of the intervention. Example questions include: What would improve the growth path or listener training for you?

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, PhD, Principal Investigator — International Psychoanalytic University Berlin
Locations (1):
- International Psychoanalytic University Berlin, Berlin, Brandenburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersson G. Internet interventions: Past, present and future. Internet Interv. 2018 Apr 6;12:181-188. doi: 10.1016/j.invent.2018.03.008. eCollection 2018 Jun. PMID 30135782
- [Background] Baumel A, Tinkelman A, Mathur N, Kane JM. Digital Peer-Support Platform (7Cups) as an Adjunct Treatment for Women With Postpartum Depression: Feasibility, Acceptability, and Preliminary Efficacy Study. JMIR Mhealth Uhealth. 2018 Feb 13;6(2):e38. doi: 10.2196/mhealth.9482. PMID 29439944
- [Background] Cornelius BL, Groothoff JW, van der Klink JJ, Brouwer S. The performance of the K10, K6 and GHQ-12 to screen for present state DSM-IV disorders among disability claimants. BMC Public Health. 2013 Feb 12;13:128. doi: 10.1186/1471-2458-13-128. PMID 23402478
- [Background] Cuijpers P, Noma H, Karyotaki E, Cipriani A, Furukawa TA. Effectiveness and Acceptability of Cognitive Behavior Therapy Delivery Formats in Adults With Depression: A Network Meta-analysis. JAMA Psychiatry. 2019 Jul 1;76(7):700-707. doi: 10.1001/jamapsychiatry.2019.0268. PMID 30994877
- [Background] Fairburn CG, Patel V. The impact of digital technology on psychological treatments and their dissemination. Behav Res Ther. 2017 Jan;88:19-25. doi: 10.1016/j.brat.2016.08.012. PMID 28110672
- [Background] Finstad K. The usability metric for user experience. Interacting with computers. 2010; 22(5): 323-327. doi: 10.1016/j.intcom.2010.04.004
- [Background] Ghani MA, Brown SE, Khan F, Wickersham JA, Lim SH, Dhaliwal SK, Kamarulzaman A, Altice FL. An exploratory qualitative assessment of self-reported treatment outcomes and satisfaction among patients accessing an innovative voluntary drug treatment centre in Malaysia. Int J Drug Policy. 2015 Feb;26(2):175-82. doi: 10.1016/j.drugpo.2014.10.002. Epub 2014 Oct 28. PMID 25577322
- [Background] Institut für Qualität und Wirtschaftlichkeit im Gesundheitswesen (IQWiG). (24.05.2017). Bericht Nr. 513, Systemische Therapie bei Erwachsenen als Psychotherapieverfahren, Abschlussbericht, Auftrag N14-02, Version 1.0; https://www.iqwig.de/download/n14-02_abschlussbericht_systemische-therapie-bei-erwachsenen_v1-0.pdf(accessed 01.09.2021)
- [Background] Johnsen AT, Petersen MA, Pedersen L, Groenvold M. Development and initial validation of the Three-Levels-of-Needs Questionnaire for self-assessment of palliative needs in patients with cancer. J Pain Symptom Manage. 2011 Jun;41(6):1025-39. doi: 10.1016/j.jpainsymman.2010.08.013. Epub 2011 Feb 9. PMID 21306865
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Karyotaki E, van Ballegooijen W. Digital self-help interventions for suicidal ideation and behaviour. Lancet Digit Health. 2020 Jan;2(1):e4-e5. doi: 10.1016/S2589-7500(19)30215-8. Epub 2019 Nov 29. No abstract available. PMID 33328038
- [Background] Kessler RC, Andrews G, Colpe LJ, Hiripi E, Mroczek DK, Normand SL, Walters EE, Zaslavsky AM. Short screening scales to monitor population prevalences and trends in non-specific psychological distress. Psychol Med. 2002 Aug;32(6):959-76. doi: 10.1017/s0033291702006074. PMID 12214795
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Messner, E. M., & Feikes, K. I. (2021). Systemische Therapie goes online. Psychotherapeut, 66, 501-510. https://doi.org/10.1007/s00278-021-00544-z
- [Background] Naslund JA, Shidhaye R, Patel V. Digital Technology for Building Capacity of Nonspecialist Health Workers for Task Sharing and Scaling Up Mental Health Care Globally. Harv Rev Psychiatry. 2019 May/Jun;27(3):181-192. doi: 10.1097/HRP.0000000000000217. PMID 30958400
- [Background] Pauley D, Cuijpers P, Papola D, Miguel C, Karyotaki E. Two decades of digital interventions for anxiety disorders: a systematic review and meta-analysis of treatment effectiveness. Psychol Med. 2023 Jan;53(2):567-579. doi: 10.1017/S0033291721001999. Epub 2021 May 28. PMID 34047264
- [Background] Revicki DA. Patient assessment of treatment satisfaction: methods and practical issues. Gut. 2004 May;53 Suppl 4(Suppl 4):iv40-4. doi: 10.1136/gut.2003.034322. PMID 15082613
- [Background] Sin J, Galeazzi G, McGregor E, Collom J, Taylor A, Barrett B, Lawrence V, Henderson C. Digital Interventions for Screening and Treating Common Mental Disorders or Symptoms of Common Mental Illness in Adults: Systematic Review and Meta-analysis. J Med Internet Res. 2020 Sep 2;22(9):e20581. doi: 10.2196/20581. PMID 32876577
- [Background] Steyer, R., Schwenkmezger, P., Notz, P. und Eid, M. (1997). Der Mehrdimensionale Befindlichkeitsfragebogen (MDBF). Göttingen: Hogrefe.
- [Background] Torok M, Han J, Baker S, Werner-Seidler A, Wong I, Larsen ME, Christensen H. Suicide prevention using self-guided digital interventions: a systematic review and meta-analysis of randomised controlled trials. Lancet Digit Health. 2020 Jan;2(1):e25-e36. doi: 10.1016/S2589-7500(19)30199-2. Epub 2019 Nov 29. PMID 33328037
- [Background] Warttig SL, Forshaw MJ, South J, White AK. New, normative, English-sample data for the Short Form Perceived Stress Scale (PSS-4). J Health Psychol. 2013 Dec;18(12):1617-28. doi: 10.1177/1359105313508346. Epub 2013 Oct 22. PMID 24155195
- [Derived] Erasmus P, Borrmann M, Ali AT, Herta S, Becker J, Moriarty G, Meinlschmidt G. Systemic therapy informed self-help and paraprofessional training in a naturalistic setting: study protocol of a digital randomised trial. Arch Public Health. 2025 May 6;83(1):119. doi: 10.1186/s13690-025-01597-1. PMID 40329383